CLINICAL TRIAL: NCT01653080
Title: Dynamic Contrast Enhanced Magnetic Resonance Imaging for Non-Invasive Diagnostic Work-Up in Solid Tumors of the Eye and Orbit.
Brief Title: MRI in Diagnosing Solid Tumors of the Eye and Orbit
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Michael V Knopp MD PhD, Principal Investigator, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OSU-0361; NCI-2012-00957 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Eye Cancer
Keywords: Solid Tumor; Eye; Orbit
MeSH Terms: conditions — Eye Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Dynamic contrast-enhanced MRI (Experimental): Patients undergo Dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI)
  Interventions: Procedure: dynamic contrast-enhanced MRI

INTERVENTIONS:
Procedure: dynamic contrast-enhanced MRI — Studies will be performed on standard clinical MR Systems which are available on Campus. With the proposed imaging technique, we are able to acquire a 3D volume covering the orbit with a temporal resolution of approximately 15s. The affected eye will be immobilized to reduce motion artifacts. A routinely used MR contrast agent will be administered in a dose of 0.1mmol/kg bodyweight.
  Other Names: DCE-MRI; Dynamic Contrast Enhanced; Magnetic Resonance Imaging

SUMMARY:
This study is being done due to a new imaging method that may help others in the future to improve evaluation of diseases in the eye and eye socket and to help make a decision concerning best treatment of the disease. Previous studies suggests that dynamic contrast enhanced MRI is ideally suited to show small structures in the eye and eye socket as well as to provide information about the eye socket such as blood circulation. This research may also provide information about the likelihood of the tumor spreading from the eye into other organs as well as correlate the study images with all other clinical imaging

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of DCE-MRI (dynamic contrast enhanced magnetic resonance imaging) as non-invasive imaging tool to image contrast enhancement in ocular and orbital tumors.

II. To compare contrast enhancement and its distribution within orbital tissue. III. To assess potential differences in contrast enhancement which help to characterize malignant lesions as well as discriminate these from benign tissue.

IV. To compare image characteristics between clinical high field end ex-vivo ultra high field magnetic resonance (MR) imaging.

V. To correlate imaging findings with obtained histology by comparing contrast enhancement parameters, e.g. maximum signal intensity, to histology characteristics, e.g. vascular density.

OUTLINE:

Patients undergo DCE-MRI.

After completion of study treatment, patients are followed up every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* The patient has an orbital mass which needs further diagnostic evaluation before treatment or for monitoring
* Able to give informed consent
* Return for follow-up visits

Exclusion Criteria:

* Patients with a lesion < 2 mm
* The patient should not participate in this study is any of the following applies to the patient: the patients has a pacemaker, metallic cardiac valve(s), magnetic material such as surgical clips, implanted electronic infusion pumps or any other condition that would interfere with the MRI, the patient has a stent somewhere in the body, the patient has a history of allergic reaction to any metals, contrast agents, x-ray dyes, the patient has claustrophobia
* Patients cannot be pregnant and prisoners will not be considered for the study
* Exposure to gadolinium-based contrast agents increases the risk for nephrogenic systemic fibrosis (NSF) in patients with acute or severe renal dysfunction; therefore, patients with the following conditions are excluded from the study:

  * Acute or chronic severe renal insufficiency (glomerular filtration rate < 30 mL/min/1.73 m^2)
  * Acute renal dysfunction due to the hepato-renal syndrome or in the perioperative liver transplantation period
* In order to identify subjects at risk for the development of NSF, the American College of Radiology (http://acr.org) recommends obtaining a medical history and a glomerular filtration rate (GFR) assessment within six weeks of MR imaging in the following patients:

  * Renal disease (including solitary kidney, renal transplant, renal tumor)
  * Age > 60
  * History of hypertension
  * History of diabetes
  * History of severe hepatic disease/liver transplant/pending liver transplant
* All subjects providing written informed consent will complete the subject history and screening form prior to MR imaging; the form will be reviewed to determine whether the subject is at risk as defined above and the availability of an estimated glomerular filtration rate (eGFR) within six weeks of anticipated MR imaging; an eGFR result greater than six weeks prior to the MRI imaging date will be repeated and evaluated for renal function; subjects with an eGFR of < 30 mL/min/1.73 m^2 will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-05-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of benign vs. malignant lesions using DCE-MRI | Up to 5 years
  Crude comparisons between the groups of patients (benign vs. malignant) will be performed using a one-way ANOVA or nonparametric Wilcoxon Rank Sum test, where appropriate. Outliers and influential covariate patterns will be identified using diagnostic plots. Depending on the complexity of the models, exact methods may be necessary.
Improved characterization of different malignant tumor types | Up to 5 years
  Logistic regression models will be applied to determine the factors most predictive of malignancy using forward selection methods described in Hosmer-Lemeshow goodness-of-fit test as well as the area under the Receiver-Operator Characteristic (ROC) curve. Outliers and influential covariate patterns will be identified using diagnostic plots. Depending on the complexity of the models, exact methods may be necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Knopp, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu